CLINICAL TRIAL: NCT02369445
Title: Investigation of Teacher-Mediated Toilet Training Using a Manualized Moisture Alarm Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Nationwide Children's Hospital (Other); Vanderbilt University (Other)
Responsible Party: Principal Investigator, Daniel Mruzek, Associate Professor of Pediatrics, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1 R40 MC27705-01-00
Record Dates: First submitted 2015-02-16; First posted 2015-02-24 (Estimated); Last update posted 2018-11-21 (Actual); Status verified 2017-10

CONDITIONS: Autistic Disorder; Enuresis
MeSH Terms: conditions — Autistic Disorder; Enuresis | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Moisture Pager (MP) Intervention Group (Experimental): This group receives the innovative toilet training intervention comprised of a wireless moisture pager (i.e., an app based on an iPod that "communicates" via electronic signal with a disposable moisture sensor located in the child's underwear).
  Interventions: Behavioral: Moisture Pager Intervention for Toilet Training
- Standard Behavioral Intervention Group (Active Comparator): This group receives standard-of-care intervention as presented in the Autism Treatment Network's Toilet Training Tool Kit (https://www.autismspeaks.org/site-wide/atn-tool-kits).
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: Moisture Pager Intervention for Toilet Training
  Arms: Moisture Pager (MP) Intervention Group
Behavioral: Standard of Care
  Arms: Standard Behavioral Intervention Group

SUMMARY:
The purpose of this pilot study is to compare an innovative toilet training strategy with a standard behavioral intervention in children with autism spectrum disorder (ASD), as implemented by teachers in the school setting. Thirty classrooms with a total of 60 children with ASD (aged 3 - 10 years) will be enrolled in the study. Each classroom will be randomly assigned to either the innovative strategy group or the standard behavioral group. The innovative strategy employs an electronic moisture pager that sends a signal when the child begins having a urine accident. Outcome measures include rate of urine accidents and rate of toilet use in the two groups.

DETAILED DESCRIPTION:
The goals of this proposed study is to develop a teacher-mediated model of toileting instruction for children with ASD in school settings that incorporates our innovative manualized moisture pager intervention (i.e., the MP intervention) and conduct a randomized controlled trial (RCT) to compare the efficacy of the MP intervention with a standard behavioral treatment (SBT).

The specific aims and related hypotheses of this proposed study are:

Aim 1: To prepare the teacher-mediated moisture pager (MP) intervention for large-scale testing in classroom settings by modifying the current parent manual for classroom use and evaluating the feasibility of the study protocol.

Hypothesis 1. The study protocol will be feasible, as indicated by achievement of recruitment targets, successful randomization, and 80% retention of both participating classroom staff and children with ASD with complete data collection.

Hypothesis 2. Teachers will deliver MP and standard behavioral treatment (SBT) intervention with >80% fidelity (as rated from teacher training fidelity checklists), and teachers in the MP and SBT intervention groups will adhere to the intervention with >80% fidelity (as rated from treatment fidelity checklists).

Hypothesis 3. Teachers participating in the MP group will report greater satisfaction with MP toilet training experience than teachers participating in the SBT group, based on teacher satisfaction surveys.

Aim 2: To compare the efficacy of the MP intervention and SBT by conducting an RCT (N= 30 classrooms with a total of 60 children with ASD aged 3 - 10 years).

Hypothesis 4. At the close of a 3-month intervention period, children in the MP group will have fewer toileting accidents and higher rate of toilet use for urination than children in the SBT group, based on data collected by teachers on pen-and-paper toileting data logs.

Hypothesis 5. At 3 months following the close of intervention, teachers in the MP group will report fewer toileting accidents and a higher rate of toileting success than children in the SBT group, as indicated through completion of toileting data logs for 3 consecutive days.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for participating children are as follows:

1. ASD diagnosis confirmed through administration of the ADOS-2,
2. status consistent with DSM-5 diagnosis of primary daytime enuresis, with the exception of DSM-5 criterion that child is at least 5 years old, confirmed by the K-SADS,
3. a positive determination of readiness for toilet training, as determined through a Toileting Readiness Checklist, developed through a review of relevant literature on toilet training children with ASD (with 4 out of 7 signs in the checklist, with 3 of these criteria required),
4. not on medication or stable for the past three months with no anticipated changes during the three-month intervention period, and
5. consent from participating teachers and parents.

Exclusion Criteria:

Exclusion criteria are:

1. medical conditions that would interfere with toilet training procedures and are not well controlled (e.g., diabetes, urinary tract infection, or seizures),
2. physical disorder that may contribute to incontinence (e.g., physical disabilities, chronic constipation) and
3. medication for enuresis.

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2014-09; Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Teacher Satisfaction with Toilet Training Experience (teacher satisfaction survey) | 60 Consecutive School Days
  A teacher satisfaction survey will be completed by each participating teacher following implementation of the intervention for 60 consecutive school days.
Number of Toileting Accidents/Day and Number of Successful Toilet Use for Urination/Day at End of Treatment (Toileting Data Logs) | 60 Consecutive School Days
  Toileting Data Logs will be completed by participating teachers during 3 consecutive days immediately prior to each of 4 visits with study personnel for both groups.
Number of Toileting Accidents/Day and Number of Successful Toilet Use (3-Month Follow-Up) (Toileting Data Logs) | Collected 3 Calendar Months After End of Intervention
  Toileting Data Logs will be completed by participating teachers during 3 consecutive days immediately prior to a follow-up appointment at 3-months following close of intervention for both groups.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel W Mruzek, PhD, Principal Investigator — University of Rochester
Locations (3):
- United States (3):
  - University of Rochester Medical Center, Rochester, New York
  - Nationwide Children's Hospital, Columbus, Ohio
  - Whitney Loring, Nashville, Tennessee